CLINICAL TRIAL: NCT01094626
Title: MRI With Secretin Enhancement to Increase Conspicuity of Pancreatic Cancer
Brief Title: Secretin-enhanced Magnetic Resonance Imaging (S-MRI) for Pancreatic Cancer Detection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pharmaceutical company did not decide to renew contract
Sponsor: Elizabeth Hecht (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Hecht, Associate Professor of Clinical Radiology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAE5847
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Cancer; Intraductal Papillary Mucinous Neoplasm
Keywords: Pancreatic adenocarcinoma; Intraductal papillary mucinous neoplasm; Imaging techniques; Pancreatic surgical resection; Synthetic human secretin
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Fifteen subjects will be randomly selected to undergo S-MRI prior to surgery. These subjects would receive Secretin, administered by IV bolus injection over 1 minute followed by a 30 second saline flush.
  Interventions: Drug: Secretin
- Controls (No Intervention): Fifteen subjects will be selected as controls, undergoing MRI without secretin-enhancement and matched for age, sex, race and tumor-type.

INTERVENTIONS:
Drug: Secretin — Subjects will each undergo an S-MRI evaluation, at a dose of 0.2 ucg/kg per exam. Secretin will be administered by IV bolus injection over 1 minute followed by a 30 second saline flush. The maximum dose of secretin will be 18.5 ucg.
  Other Names: RG1068
  Arms: Experimental

SUMMARY:
The aim of the study is to evaluate the utility of secretin-enhanced MRI (S-MRI) in detecting and measuring pancreatic lesions in patients with known adenocarcinoma or Intraductal papillary mucinous neoplasm (IPMN) lesions. The hypothesis is that S-MRI is superior to MRI without secretin enhancement (N-MRI) in increasing tumor conspicuity, allowing for improved identification and more accurate measurement of lesions or precursor lesions in the pancreas.

DETAILED DESCRIPTION:
Pancreatic cancer remains the fourth leading cause of cancer-related death in the United States and is marked by advanced stage at diagnosis and a high mortality rate. Intraductal papillary mucinous neoplasm (IPMN) is a cystic lesion that can be potentially cancerous, leading to pancreatic adenocarcinoma. Currently, there is no existing imaging modality that is both sensitive and cost-effective enough in accurately measuring or detecting adenocarcinoma and IPMN. Improving the methods used in identification and localization of this disease is critical.

Secretin, a hormone produced by duodenal mucosal cells increases blood-flow to the pancreas. The investigators' hypothesis is that as secretin increases blood flow to the pancreas, there will be increased conspicuity in areas of dysplasia/cancer where there is minimal blood-flow, enhancing tumor detection. The investigators are conducting a prospective, randomized-control pilot study of thirty subjects with IPMN or pancreatic cancer who are undergoing surgical resection at Columbia University's Pancreas Center. Fifteen subjects will be randomly selected to undergo S-MRI prior to surgery and fifteen subjects will be selected as controls, undergoing MRI without secretin-enhancement and matched for age, sex, race and tumor-type. The investigators will first evaluate if secretin allows for increased tumor conspicuity, enhanced visualization of the lesion, by comparing the calculated tumor conspicuity of S-MRI to N-MRI groups.

The investigators will then assess if S-MRI imaging allows for increased accuracy in lesion measurements by looking at the concordance in measurements between S-MRI and tumor specimens post-resection as compared to the concordance in measurements between N-MRI and tumor specimens post-resection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed IPMN/pancreatic adenocarcinoma by biopsy or fine needle or suspected IPMN/pancreatic adenocarcinoma based on imaging
* Scheduled for surgical resection
* Willingness to provide informed consent.

Exclusion Criteria:

* Any contraindication to magnetic resonance imaging (MRI), including but not limited to implanted metal devices (e.g. pacemaker, berry aneurysm clips, neural stimulator or cochlear implants)
* Unresectable tumor
* Other abdominal neoplasm in addition to neoplasm in pancreas
* Contraindication to surgery, including but not limited to recent myocardial infarction (MI) (within 6 weeks) or poor pulmonary function
* History of sensitivity to secretin
* Pregnancy
* Estimated glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 (as per Modification of Diet in Renal Disease (MDRD) Study equation)
* Unwillingness or inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Difference in lesion conspicuity between S-MRI and N-MRI | 30 days
  The primary outcome is whether S-MRI allows for better tumor detection secondary to anticipated increased conspicuity of tumor due to secretin's effect on increasing blood flow to the normal pancreas as compared to N-MRI. Determining S-MRI's efficacy versus that of N-MRI will be carried out by comparing tumor conspicuity measurements in S-MRI and N-MRI groups. Tumor conspicuity will be measured by calculating the contrast to noise ratio, placing region of interest (ROI) on tumor and adjacent tissue and dividing by image noise.

SECONDARY OUTCOMES:
Concordance of tumor measurements between S-MRI images and tumor specimens post-resection vs. concordance of tumor measurements between N-MRI and tumor specimens post-resection | 45 days
  The secondary outcome will be the discrepancy in tumor size estimated from MRI and "confirmed" from post-surgical specimens. Tumor size estimated from MRI scans will be determined by measuring the greatest linear dimension (metric) of the lesion. Tumor size estimated by pathology will be directly measured using a linear scale (metric), taking the greatest linear dimension of the resected tumor. The discrepancy in estimated versus "confirmed" tumor size will be compared between S-MRI and N-MRI groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hecht, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No